CLINICAL TRIAL: NCT00240591
Title: A MULTI-CENTER LONG-TERM FOLLOW-UP STUDY OF PATIENTS WITH LOW-GRADE NON-HODGKIN'S LYMPHOMA PREVIOUSLY TREATED WITH TOSITUMOMAB AND/OR IODINE I 131 TOSITUMOMAB IN STUDIES RIT-I-000, RIT-II-001, RIT-II-002, RIT-II-004, or CP-97-012
Brief Title: Patients With Low-Grade Non-Hodgkin's Lymphoma Previously Treated With Tositumomab and/or Iodine I 131 Tositumomab
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: BEX104526
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: BEXXAR; Tositumomab; Iodine I 131 Tositumomab; low-grade follicular lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study for the long-term follow-up of patients who completed at least two years of follow-up after treatment with Tositumomab and/or Iodine I 131 Tositumomab (BEXXAR)on Study RIT-I-000, RIT-II-001, RIT-II-002, RIT-II-004 or CP-97-012. All patients will be assessed for survival and disease status, including subsequent therapy for NHL, and for long term safety. Laboratory evaluations consisting of a TSH level (for all patients) and a complete blood cell (CBC) count with a differential and platelet count (for patients in continuing response only) will be obtained annually through Year 10 post treatment with Tositumomab and/or Iodine I 131 Tositumomab.

Patients that remain in response to their previous treatment with BEXXAR, will additionally be followed radiographically for response and progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have enrolled in one of the following Corixa sponsored clinical trials: RIT-I-000, RIT-II-001, RIT-II-002, RIT II-004 or CP-97-012 and are >2 years post Tositumomab and/or Iodine I 131 Tositumomab administration.
* Patients must give written informed consent by signing an IRB/ethics committee approved consent form prior to entry on this follow-up study.

Exclusion Criteria:

* Inability to meet the above referenced inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with NHL previously treated at least 2 years ago with Tositumomab and/or Iodine I 131 Tositumomab on Study RIT-I-000, RIT-II-001, RIT-II-002, RIT-II-004, or CP-97-012.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2003-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
None - Administrative non interventional study to obtain long term safety and efficacy data. | Subjects enrolled in Study BEX104526 were followed for continued response (as applicable) and safety every 6 months for Years 3 through 5 post-treatment with TST/I-131 TST. Beginning at Year 6, subjects were assessed annually through Year 10 inclusive.
  Study BEX104526 (formerly Corixa Study CCBX001-051) was designed to obtain long-term safety and efficacy data from the surviving subjects who completed at least 2 years of follow-up following administration of TST/I-131 TST while on Study BEX104728 (RIT-I-000), BEX104731 (RIT-II-001), BEX104504 (RIT-II-004), BEX104515 (RIT-II-002), or BEX104507 (CP-97-012). Analyses will be performed according to one of the five primary interventional protocols.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline